CLINICAL TRIAL: NCT06184347
Title: A Prospective and Observational Investigation on Chronic Hepatitis B Virus Infection and Related Liver Diseases Via Systematic Screening in General Population
Brief Title: Population-wide Research for HBV-related Liver Diseases in Maoming City
Acronym: PreMAO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2023-474
Record Dates: First submitted 2023-12-13; First posted 2023-12-28 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: HBV Infection; Chronic Hepatitis B; Cirrhosis; HCC
MeSH Terms: conditions — Hepatitis B, Chronic; Fibrosis | interventions — Hepatitis B Surface Antigens

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Screening group: All participants will receive an HBsAg finger blood test and a questionnaire gathering their personal information and medical history concerning viral hepatitis, cirrhosis, and hepatocellular carcinoma. Individuals positive for HBsAg will undergo further clinical detections to distinguish dormant liver diseases and HCC.
  Interventions: Other: Rapid tests for HBsAg
- Control group: All subjects in this arm will be followed by linkage to the Guangdong Provincial Center for Disease Control and Prevention, Cancer Registry, and Population Registry.

INTERVENTIONS:
Other: Rapid tests for HBsAg — Participants in the screening group will firstly receive the HBsAg screening using a finger blood test.
  The laboratory examination includes blood routine test (white blood cell count [WBC], red blood cell count [RBC], hemoglobin [HGB], platelet count [PLT]), liver function (total bilirubin [TBIL], albumin [ALB], alanine aminotransferase [ALT]), HBV serologic markers, alpha-fetoprotein(AFP) , abnormal Prothrombin II (PIVKA II) and HBV-DNA.
  The imaging examination includes liver ultrasound, abdominal CT, or MRI. HBsAg-positive participants also undergo liver ultrasound examination. If suspicious liver nodules or elevated AFP levels are detected, further refinement through abdominal CT or MRI is recommended.
  Other Names: Laboratory examination of sample of blood; Imaging examination
  Groups: Screening group

SUMMARY:
Hepatitis B virus (HBV) infection is a major public health problem and chronic HBV infection affects about 296 million people worldwide and is the leading etiology of cirrhosis and hepatocellular carcinoma globally. China takes up a great deal of the responsibility towards the goal of "eliminating viral hepatitis by 2030" released by the World Health Organization (WHO), as China has the world's largest burden of HBV infection. The current diagnostic rate barely reaches 24%, which is significantly short of the target diagnostic rate of 90% proposed by WHO. Progression from chronic hepatitis B (CHB) to hepatic complications-fibrosis, cirrhosis, and HCC-can be prevented significantly by preemptive antiviral therapy. However, the onset of CHB seldom manifests with typical symptoms, and most cases at their first diagnosis have progressed to end-stage liver diseases. Therefore, early detection of CHB and its complications that not only raises public awareness of preventing infection but also brings the patients into the management system is urgent blocking the progression to cirrhosis and HCC.

The study is a prospective and observational study involving community-based screening of chronic HBV infection and related liver diseases systematically among the general population of Guangdong Province, China. Individuals in Maoming City, aged 20-70 years, will be enrolled in the screening group for the HBsAg screening using a finger blood test. Positive participants will receive further examinations including laboratory and imaging examinations to discover HBV-related liver diseases. The control group will be enrolled from the general population in two similar cities.

By thoroughly investigating the epidemiological landscape and antiviral situation of chronic hepatitis B through population screening, this study intends to furnish the administration with updated epidemiological data. Additionally, the project seeks to establish a CHB screening cohort to enhance early diagnosis and treatment rates for both HBV-related liver diseases. Collectively, the study aspires to improve the overall prognosis for patients with chronic HBV infection, reduce CHB-related mortality, and ultimately put forward valuable healthcare insights and evidence-based medicine (EBM) practices for the effective implementation of CHB screening and management.

DETAILED DESCRIPTION:
Sample selection Individuals aged from 20-70 years old who permanently reside in Maoming City will be enrolled in the screening group.

The natural population from another two cities which share economic, climatic, and customary similarities with Maoming City will be enrolled in the control group.

Participants recruitment Participants who voluntarily attend the screening project will be recruited to the screening group. Personal and medical information of the control group will be fetched from the Guangdong Provincial Center for Disease Control and Prevention, the Cancer Register, the Population Register, and other relevant systems.

Informed consent Informed consent forms will be collected at the recruitment in the screening group.

Questionnaires Questionnaires will be conducted face-to-face by well-trained investigators to gather the personal information of the participants in the screening group and inquire about the previous and current medical history of them and their families concerning viral hepatitis, cirrhosis, and HCC.

HBsAg screening test Participants in the screening group will firstly receive the HBsAg screening using a finger blood test.

Laboratory and imaging examinations Participants positive for the HBsAg screening test in the screening group will undergo further clinical examination to determine if their infections have developed CHB and even HCC. The laboratory examination includes blood routine tests (white blood cell count [WBC], red blood cell count [RBC], hemoglobin [HGB], platelet count [PLT]), liver function (total bilirubin [TBIL], albumin [ALB], alanine aminotransferase [ALT]), HBV serologic markers, alpha-fetoprotein (AFP), abnormal Prothrombin II (PIVKA II) and HBV-DNA. Patients with HBsAg-positive status undergo liver ultrasound examination. If suspicious liver nodules or elevated AFP levels are detected, further refinement through abdominal CT or MRI is recommended.

ELIGIBILITY:
Inclusion Criteria:

1. Screening Group

   Individuals with all the following characteristics can be included:
   1. Aged from 20 to 70;
   2. From the residential population of Maoming City, Guangdong Province;
   3. Voluntarily participate and provide written informed consent forms.
2. Control Group

Individuals with all the following characteristics can be included:

1. Aged from 20 to 70;
2. From the residential population of Wuchuan City and Yangchun City, Guangdong Province.

Exclusion criteria:

1. Screening Group

   Individuals with all the following characteristics should be excluded:
   1. Floating population and temporary residents;
   2. Diagnosed with severe mental diseases who are unable to communicate normally;
   3. Determined by the researchers to be unsuitable for this study;
2. Control Group The control group data will be collected and organized through relevant systems such as the Guangdong Provincial Center for Disease Control and Prevention, the Cancer Register, and the Population Register, requiring no exclusion.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population in Guangdong Province
Sampling Method: Non-Probability Sample
Enrollment: 3700000 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Estimation of the HBV-related liver disease incidences in Guangdong Province | 2024.02-2025.08
  The incidences of HBV-related liver diseases will be calculated as the percentage of patients diagnosed with Hepatitis B, cirrhosis, and HCC in the screening and control groups, which will be used to estimate the HBV-related liver disease incidences in Guangdong Province.
Propotion of participants who are eligible for and would benefit from antiviral therapy. | 2024.02-2025.08
  Propotion of participants who are eligible for and would benefit from antiviral therapy will be based on the percentage of patients who need antiviral therapy after being diagnosed with Hepatitis B, cirrhosis, and HCC in the screening group.

SECONDARY OUTCOMES:
Estimation of the Hepatitis B virus infection rate in Guangdong Province | 2024.02-2025.08
  The Hepatitis B virus infection rate will be based on the percentage of subjects positive for HBV in the screening and control groups, which will be used to estimate the Hepatitis B virus infection rate in Guangdong Province.
Early diagnosis rate of liver cirrhosis or hepatocellular carcinoma | 2024.02-2025.08
  The early diagnosis rate of liver cirrhosis and hepatocellular carcinoma is based on the percentage of CHB patients who have received a confirmed diagnosis of cirrhosis or HCC by the total number of individuals with CHB in the screening group.
The current therapeutic rate of chronic hepatitis B | 2024.02-2025.08
  The current therapeutic coverage of chronic hepatitis B will be based on the percentage of patients who accepted antiviral therapy after being diagnosed with HBV infection before screening.

CONTACTS AND LOCATIONS:
Overall Officials: Li Liu, Principal Investigator — Nanfang Hospital, Southern Medical University

REFERENCES:
- [Background] Jeng WJ, Papatheodoridis GV, Lok ASF. Hepatitis B. Lancet. 2023 Mar 25;401(10381):1039-1052. doi: 10.1016/S0140-6736(22)01468-4. Epub 2023 Feb 9. PMID 36774930
- [Background] Liu Z, Lin C, Mao X, Guo C, Suo C, Zhu D, Jiang W, Li Y, Fan J, Song C, Zhang T, Jin L, De Martel C, Clifford GM, Chen X. Changing prevalence of chronic hepatitis B virus infection in China between 1973 and 2021: a systematic literature review and meta-analysis of 3740 studies and 231 million people. Gut. 2023 Nov 24;72(12):2354-2363. doi: 10.1136/gutjnl-2023-330691. PMID 37798085
- [Background] Su S, Wong WC, Zou Z, Cheng DD, Ong JJ, Chan P, Ji F, Yuen MF, Zhuang G, Seto WK, Zhang L. Cost-effectiveness of universal screening for chronic hepatitis B virus infection in China: an economic evaluation. Lancet Glob Health. 2022 Feb;10(2):e278-e287. doi: 10.1016/S2214-109X(21)00517-9. PMID 35063115
- [Background] Hsu YC, Huang DQ, Nguyen MH. Global burden of hepatitis B virus: current status, missed opportunities and a call for action. Nat Rev Gastroenterol Hepatol. 2023 Aug;20(8):524-537. doi: 10.1038/s41575-023-00760-9. Epub 2023 Apr 6. PMID 37024566
- See also: HBV progress towards coverage targets — https://cdafound.org/polaris-countries-dashboard/